CLINICAL TRIAL: NCT04834713
Title: Study on the Relationship Between Neutrophil-mediated Thrombocytopenia and the Condition and the Course of Disease in Patients With HFRS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2020-013
Record Dates: First submitted 2020-12-24; First posted 2021-04-08 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Hemorrhagic Fever With Renal Syndrome
MeSH Terms: conditions — Hemorrhagic Fever with Renal Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Mild patients: defined as patients who had kidney injury without oliguria and hypotension
  Interventions: Other: clinical classification of HFRS
- moderate patients: defined as patients who had uremia, effusion (bulbar conjunctiva), hypotension, hemorrhage (skin and mucous membranes), and AKI with typical oliguria
  Interventions: Other: clinical classification of HFRS
- severe patients: defined as patients who had severe uremia, effusion (bulbar conjunctiva and either peritoneum or pleura), hemorrhage (skin and mucous membranes), hypotension and AKI with oliguria (urine output of 50-500 mL/day) for ≤ 5 days or anuria (urine output of < 100 mL/day) for ≤ 2 days
  Interventions: Other: clinical classification of HFRS
- critical patients: defined as patients who usually had one or more of the following complications compared with the severe patients: refractory shock (≥ 2 days), visceral hemorrhage, heart failure, pulmonary edema, brain edema, severe secondary infection, and severe AKI with oliguria (urine output of 50-500 mL/day) for > 5 days or anuria (urine output of < 100 mL/day) for > 2 days
  Interventions: Other: clinical classification of HFRS
- healthy control: defined as people without HFRS

INTERVENTIONS:
Other: clinical classification of HFRS — Based upon clinical classification of HFRS , the patients were classified into four types
  Groups: Mild patients; critical patients; moderate patients; severe patients

SUMMARY:
Thrombocytopenia is an important pathological feature of HFRS（Hemorrhagic Fever With Renal Syndrome, HFRS）. However, the cause of thrombocytopenia in HFRS is not yet fully understood. Neutrophils, as the largest number of white blood cells in the human body, can widely participate in the immune process of viral infections. Previous studies have found that the neutrophils of patients with acute myocardial infarction can interact with activated platelets and further mediate platelet phagocytosis.Therefore, this study aims to systematically elucidate the immunological process of neutrophil mediated thrombocytopenia in patients with HFRS by exploring the correlation between platelet activation, neutrophil activation and neutrophil proportion of adherent / phagocytic platelets peripheral blood of HFRS patients, and to analyze its relationship with the course of HFRS disease, which lays a theoretical foundation for further understanding the pathogenesis of HFRS and provides a basis for clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Clinical diagnosis meets the diagnostic criteria of the national HFRS prevention and treatment plan (Hantavirus-specific IgM antibody is positive). The classification and staging standards of HFRS patients are based on the "Expert Consensus of Shaanxi Province on Diagnosis and Treatment of Hemorrhagic Fever with Renal Syndrome".

Exclusion Criteria:

* Age <18 years;
* Have a history of kidney disease;
* Have a history of liver disease;
* Have a history of malignant tumor;
* Receive dialysis treatment before admission;
* Combined with hypertension, coronary heart disease and diabetes history;
* Combined with HIV infection and patients with autoimmune diseases and pregnancy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This project intends to collect about 160 inpatients (the First Affiliated Hospital of Xi'an Jiaotong University) who were diagnosed with HFRS between 2021.01-2023.06 for follow-up research, including about 40 cases of light, medium, severe, and critical. 40 healthy people served as normal controls.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Changes in the platelet activation ratio, % | through study completion, an average of 2 year
  flow cytometry
Changes in neutrophils MPO content, MFI | through study completion, an average of 2 year
  enzyme-linked immunosorbent assay
Changes in the neutrophils with adherent platelets, % | through study completion, an average of 2 year
  flow cytometry
Changes in the neutrophils with internalized platelets, % | through study completion, an average of 2 year
  flow cytometry

SECONDARY OUTCOMES:
Changes in Neutrophils Mac-1 expression, MFI | through study completion, an average of 2 year
  flow cytometry
Changes in the platelets with phosphatidylserine exposure,% | through study completion, an average of 2 year
  flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: xiaojiao Li, Study Director — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong university, Xi'an, Shaanxi, China